CLINICAL TRIAL: NCT07146308
Title: Multiscale Causal Disease Warning and Assisted Diagnosis: Multi-omics Mechanisms of Lifestyle Intervention in Regulating Blood Glucose
Brief Title: Multi-omics Mechanisms of Lifestyle Intervention in Regulating Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Huating, Professor, Shanghai 6th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-KY-239(K)
Record Dates: First submitted 2025-07-13; First posted 2025-08-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle intervention Arm (Experimental)
  Interventions: Other: Lifestyle Management

INTERVENTIONS:
Other: Lifestyle Management — Participants will undergo dietary and exercise interventions. The dietary intervention includes breakfast, lunch, and dinner, while the exercise intervention consists of both aerobic and resistance training.

SUMMARY:
The mechanisms by which lifestyle interventions regulate blood glucose remain incompletely understood. Traditional research has predominantly focused on single targets or pathways, making it difficult to comprehensively elucidate the complex biological regulatory networks. This study systematically investigates the effects of lifestyle interventions on blood glucose and explores their molecular mechanisms. Through integrated multi-omics analysis-including genomics, proteomics, metabolomics, and microbiomics-investigators aim to identify key biological pathways and molecular targets through which dietary, exercise, and other lifestyle interventions influence glucose regulation, as well as discover biomarkers that reflect the efficacy of these interventions. Building upon these findings, investigators will establish a multi-omics molecular network model linking lifestyle interventions to glucose regulation and develop an auxiliary decision-making system for personalised diabetes diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years

Exclusion Criteria:

* Severe chronic diabetic complications or recent acute diabetic complications
* Type 1 diabetes mellitus
* Early-onset diabetes
* Patients currently using insulin therapy
* Recent severe hypoglycemic episodes
* Secondary obesity
* Pregnancy, severe hepatic/renal diseases, thyroid disorders, acute infections, psychiatric disorders, or other conditions that may interfere with study outcomes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-08-31 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Post-intervention incremental area under the glucose curve (iAUC) measured by continuous glucose monitoring (CGM) | 4 weeks

SECONDARY OUTCOMES:
Time in Range (TIR), Time Above Range (TAR), Time Below Range (TBR) Measured by Continuous Glucose Monitoring | Baseline and 4 weeks
Composite glucose metabolism profile | Baseline and 4 weeks
  A composite outcome summarizing glucose metabolism indicators, including:
  HbA1c (%), Fasting plasma glucose (mmol/L), 60- and 120-minute plasma glucose during OGTT (mmol/L), Fasting and post-load insulin (μU/mL), Fasting and post-load C-peptide (ng/mL), Homeostatic Model Assessment of Insulin Resistance (HOMA-IR, index), etc.
Composite kidney function profile | Baseline and 4 weeks
  A composite outcome summarizing kidney function indicators, including:
  Serum creatinine (mg/dL), Blood urea nitrogen (mg/dL), Estimated glomerular filtration rate (eGFR, mL/min/1.73m²), etc.
Composite liver function profile | Baseline and 4 weeks
  A composite outcome summarizing liver function biomarkers, including: Alanine aminotransferase (ALT, U/L), Aspartate aminotransferase (AST, U/L), Gamma-glutamyl transferase (GGT, U/L), Alkaline phosphatase (ALP, U/L), Total bilirubin (μmol/L), Albumin (g/L), etc.
Lipid profile | Baseline and 4 weeks
  Total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides, etc.
Inflammatory markers | Baseline and 4 weeks
  High-sensitivity C-reactive protein, etc.
Retinopathy status (digital retinal fundus imaging) | Baseline and 4 weeks
  Retinopathy grading assessed by standardized digital retinal fundus images.
Composite dietary intake profile | At each meal, aggregated dayly, up to 28 days
  A composite outcome summarizing dietary intake indicators, including:
  Total daily energy intake (kcal), Macronutrient distribution and intake (percentage and intake (gram) of total energy from carbohydrate, protein, fat, etc.), Selected micronutrient intakes (mg/day), etc.
Composite physiological monitoring profile from wearables | Daily measurements, up to 28 days
  This composite outcome includes multiple physiological parameters measured via wearable devices to assess rest and recovery status. The parameters include: Sleep duration (hours), Sleep stages (percent time in REM, deep, light), Respiratory rate (breaths per minute), Heart rate (n per minute), Other relevant physiologic signals (as available from device).
Lifestyle management-related parameters | Baseline and 4 weeks
  A structured lifestyle management questionnaire will be administered to assess multiple aspects of participants' personal health-related behaviours and preferences. This includes: food preference, exercise preference, past medical histories, health-related personal behaviours, etc.
Complete Blood Count | Baseline and 4 weeks
Routine urine test | Baseline and 4 weeks
Mean Glucose measured by continuous glucose monitoring | Baseline and 4 weeks
Glucose Variability measured by continuous glucose monitoring | Baseline and 4 weeks
Area Under the Curve (AUC) measured by continuous glucose monitoring | Baseline and 4 weeks
Body weight | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Body weight measured in kilograms using a calibrated digital scale.
Height | Baseline
  Standing height measured in meters using a stadiometer.
BMI | Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
  Calculated as weight in kilograms divided by height in meters squared (kg/m²).
Waist, hip and thigh circumference | Baseline, 4 weeks
  Measured in centimeters
Systolic and Diastolic Blood Pressure | Baseline, 4 weeks
  Systolic and diastolic blood pressure will be measured in millimeters of mercury (mmHg) using an automated sphygmomanometer. Participants will be seated quietly for at least 5 minutes before measurement, and two readings will be taken 1-2 minutes apart; the average will be recorded.
Resting heart rate | Baseline, 4 weeks
  Resting heart rate will be measured in beats per minute (bpm) using the automated sphygmomanometer's pulse reading or a validated heart rate monitor. Measurements will be taken in the seated position after at least 5 minutes of rest.
Genomic profiling | Baseline and 4 weeks
  Whole-genome sequencing for variant analysis.
Metabolomics profiling | Baseline and 4 weeks
  Untargeted metabolomics profiling using LC-MS/MS.
Proteomics profiling | Baseline and 4 weeks
  Quantitative proteomics using mass spectrometry.
Fecal Metagenomics | Baseline and 4 weeks
  Shotgun metagenomic sequencing of fecal samples to characterize gut microbiome taxonomic composition and functional gene profiles.
Fecal Metabolomics | Baseline and 4 weeks
  Untargeted metabolomics profiling of fecal samples using liquid chromatography-mass spectrometry (LC-MS/MS) to identify and quantify metabolites.
Lipidomics profiling | Baseline and 4 weeks
  Targeted lipidomics analysis of serum lipids using mass spectrometry to quantify lipid species and subclasses.
PBMC Multi-omics Profiling | Baseline and 4 weeks
  Peripheral blood mononuclear cells (PBMCs) will be analyzed using multiple omics platforms to comprehensively profile molecular changes. Analyses will include:
  Transcriptomics: Bulk RNA sequencing to quantify gene expression. Epigenomics: Genome-wide DNA methylation profiling using bisulfite sequencing. Phosphoproteomics: Quantitative analysis of phosphorylated proteins using mass spectrometry-based phosphoproteomics to assess signaling pathway activation.
  Single-cell Transcriptomics: Single-cell RNA sequencing to characterize cell type-specific transcriptional changes.
  Results from these platforms will be integrated to generate a composite PBMC multi-omics dataset.
Glycemic Excursions Composite Score from Continuous Glucose Monitoring | Baseline and 4 weeks
  Glycemic excursions will be evaluated using a composite measure derived from continuous glucose monitoring (CGM) data. The composite score will integrate multiple CGM-derived metrics, including:
  Mean glucose (mg/dL) Standard deviation of glucose (mg/dL) Coefficient of variation (%) Mean amplitude of glycemic excursions (MAGE, mg/dL)
Exercise heart rate | Each exercise session, aggregated daily up to 28 days
  Average heart rate during each exercise session.
Exercise frequency | Each exercise session, aggregated daily up to 28 days
  Number of completed exercise sessions.
Energy expenditure per session | Each exercise session, aggregated daily up to 28 days
  Energy expenditure estimated by wearable device.
Exercise duration | Each exercise session, aggregated daily up to 28 days
  Duration of each exercise session.
Number of sets and repetitions | Each exercise session, aggregated daily up to 28 days
  Total sets and repetitions performed during exercise.
Exercise intensity/load | Each exercise session, aggregated daily up to 28 days
  Intensity or load during exercise session (self-reported using Borg RPE scale or device-recorded).
Excess post-exercise oxygen consumption | Each exercise session, aggregated daily up to 28 days
  Post-exercise oxygen consumption recorded by wearable device.
Fat mass | Baseline, 1 week, 2 week, 3 week, 4 week
  Total fat mass measured by bioelectrical impedance analysis.
Fat-free mass | Baseline, 1 week, 2 week, 3 week, 4 week
  Fat-free mass measured by bioelectrical impedance analysis.
Body fat percentage | Baseline, 1 week, 2 week, 3 week, 4 week
  Percentage of total body weight as fat.
Visceral fat area | Baseline, 1 week, 2 week, 3 week, 4 week
  Estimated visceral fat area.
Muscle mass | Baseline, 1 week, 2 week, 3 week, 4 week
  Skeletal muscle mass measured by bioelectrical impedance analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China